CLINICAL TRIAL: NCT00385203
Title: An Open-Label, Phase II Study to Evaluate the Biological Activity of Cediranib (AZD2171) as Measured by [F 18] Fluoro 2 Deoxy D Glucose - Positron Emission Tomography (FDG-PET) Response, in Patients With Metastatic Gastro-Intestinal Stromal Tumours (GIST) Resistant or Intolerant to Imatinib Mesylate
Brief Title: The Biological Activity of Cediranib (AZD2171) in Gastro-Intestinal Stromal Tumours(GIST).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00046
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Gastrointestinal Stromal Tumors; Soft Tissue Sarcomas
Keywords: cancer; tumour; advanced cancer; Metastatic Gastro-Intestinal Stromal Tumours; gastro-intestinal cancer; RECENTIN
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma; Neoplasms | interventions — cediranib

INTERVENTIONS:
Drug: AZD2171 — 45 mg oral tablet once daily dose
  Other Names: cediranib; RECENTIN™

SUMMARY:
To determine the anti-tumour activity and biological effects of cediranib (AZD2171) at a dose of 45mg, primarily in Gastrointestinal Stromal Tumour (GIST) patients who are resistant to imatinib mesylate (current standard therapy) and also in patients with metastatic Soft Tissue Sarcoma (STS) resistant to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of GIST which is resistant or intolerant to imatinib mesylate, or metastatic STS, which is refractory to standard therapies or for which no standard therapy exists

Exclusion Criteria:

* Patients with type I insulin-dependent diabetes or poorly-controlled type II insulin-independent diabetes.
* Patients with a history of poorly controlled high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, MD, Study Director — AstraZeneca
Locations (2):
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Sutton

REFERENCES:
- [Derived] Judson I, Scurr M, Gardner K, Barquin E, Marotti M, Collins B, Young H, Jurgensmeier JM, Leahy M. Phase II study of cediranib in patients with advanced gastrointestinal stromal tumors or soft-tissue sarcoma. Clin Cancer Res. 2014 Jul 1;20(13):3603-12. doi: 10.1158/1078-0432.CCR-13-1881. Epub 2014 Apr 8. PMID 24714778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled: 45mg GIST=26, 45mg STS=10; Full analysis set: 45mg GIST=25, 45mg STS=10; Safety set: 45mg GIST=24, 45mg STS=10. 36 patients were enrolled and 35 patients were randomized. One GIST patient consented but had an adverse event and was withdrawn from the study before they were randomised.
Groups:
- Cediranib 45 mg/Day GIST: 26 Gastrointestinal Stromal tumour patients (GIST) were enrolled (informed consent received), one patient was enrolled but had an AE prior to randomisation so were withdrawn from the study. No demographic data were obtained for this patient.
- Cediranib 45 mg/Day STS: 10 Soft Tissue Sarcomas (STS) patients were randomised.
Period: Overall Study
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Started | 26 | 10
Completed | 0 | 3
Not Completed | 26 | 7
Not completed — Adverse Event | 5 | 4
Not completed — Death | 1 | 0
Not completed — Condition under investigation worsened | 18 | 3
Not completed — Incorrect enrollment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cediranib 45 mg/Day GIST: Cediranib 45 mg/Day: 25 patients with Gastrointestinal Stromal Tumour (GIST) randomised
- Cediranib 45 mg/Day STS: Cediranib 45 mg/Day: 10 patients with Soft Tissue Sarcomas (STS) randomised
- Total: Total of all reporting groups
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS | Total
Number analyzed (Participants) | 25 | 10 | 35
Age Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 56.1 (9.8) | 44.6 (9.4) | 52.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 8 | 6 | 14
    Male | 17 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Standardised Uptake Value (SUV)Max at Day 8, Central Review, (GIST) Gastrointestinal Stromal Tumours Patients.
Description: [F 18] Fluoro 2 Deoxy D Glucose - Positron Emission Tomography (FDG-PET). Tumour metabolic activity as assessed by Change in Standardised Uptake Value (SUVMax) at Day 8 (measured by central review), in Patients with GIST tumours. SUVmax at Day 8 minus SUVmax at Baseline.
Time Frame: Baseline and 8 days after dosing.
Population: As per the protocol the analysis was for GIST patients only (not STS patients). For patients to be included in the analysis they had to have scans with readable results at both timepoints (baseline and Day 8).
Measure: Mean (95% Confidence Interval); unit: g/mL
Groups:
- Cediranib 45 mg/Day STS: Cediranib 45 mg/Day patients with Soft Tissue Sarcomas (STS): 10 patients randomised and received at least one dose of treatment
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 22 | 0
g/mL | -0.515 [-1.480 to 0.450] |

2. Primary Outcome: Tumour Metabolic Activity as Assessed by Change in Central Review of Standardised Uptake Value (SUVMax) at Day 29, in Patients With GIST Tumours. SUVmax at Day 29 Minus SUVmax at Baseline.
Description: SUVmax at Day 29 minus SUVmax at baseline, based on central review, GIST patients
Time Frame: FDG-PET assessment at Baseline and 29 days after dosing.
Population: As per the protocol the analysis was for GIST patients only (not STS patients). For patients to be included in the analysis they had to have scans with readable results at both timepoints (baseline and Day 29).
Measure: Mean (95% Confidence Interval); unit: g/mL
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 20 | 0
g/mL | -0.172 [-1.380 to 1.040] |

3. Secondary Outcome: Objective Tumour Response, Investigator Review
Description: Number of patients with complete (CR) /partial response (PR) (based on RECIST) as assessed by the Investigator. CR is defined as Disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of Longest Diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: RECIST at Baseline, Weeks 8, 16 and every 12 weeks thereafter until progression.
Measure: Number; unit: Participants
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 24 | 10
Participants | 0 | 4

4. Secondary Outcome: -Tumour Activity as Measured by Major Axis (Axial Plane) at Week 8 in GIST/STS Patients by Central Review of CT Images.
Description: Central review of CT images taking the longest diameter measured in millimetres at week 8 [major axis (axial plane)] minus the longest diameter measured in millimetres at baseline.
Time Frame: CT assessments at Baseline and Week 8
Population: As per the protocol the formal statistical analysis was performed for the GIST grouppatients only, STS patients were summarised (not STS patients). For patients to be included in the analysis they had to have CT scans at both timepoints (baseline and week 8).
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 18 | 8
mm | 2.734 [-1.76 to 7.230] | -1.015 [-7.22 to 5.19]

5. Secondary Outcome: Anti-tumour Activity as Measured by Major Axis (Axial Plane) at Week 16 in GIST/STS Patients by Central Review of CT Images.
Description: Central review of CT images taking the longest diameter measured in millimetres at week 16 [major axis (axial plane)] minus the longest diameter measured in millimetres at baseline.
Time Frame: CT assessments at Baseline and Week 16.
Population: As per the protocol formal statistical analysis was performed for the GIST group only, STS patients were summarised. For patients to be included in the analysis they had to have CT scans at both timepoints (baseline and week 8).
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 13 | 5
mm | 5.028 [-1.120 to 11.180] | -8.114 [-15.74 to -0.49]

6. Secondary Outcome: Tumour Activity as Measured by Total Lesion Volume at Week 8 in GIST Patients by Central Review of CT Images.
Description: Central review of CT images taking the total lesion volume at week 8 minus the total lesion volume at baseline.
Time Frame: CT assessments at Baseline and Week 8
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: cm3
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 18 | 8
cm3 | 19889.31 [-7054.96 to 46833.58] | 5106.30 [-21840.10 to 32052.70]

7. Secondary Outcome: Anti-tumour Activity as Measured by Total Lesion Volume at Week 16 in GIST Patients by Central Review of CT Images.
Description: Central review of CT images taking the total lesion volume at week 16 minus the total lesion volume at baseline.
Time Frame: CT assessments at Baseline and Week 16
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: cm3
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Number analyzed (Participants) | 13 | 5
cm3 | 43202.54 [-4505.18 to 90910.27] | -6479.65 [-15411.92 to 2452.63]

ADVERSE EVENTS:
Description: Adverse events are reported for randomised patients who received at least one dose of treatment.
Groups:
- Cediranib 45 mg/Day GIST: Cediranib 45 mg/Day patients with Gastrointestinal Stromal Tumour (GIST): 24 patients randomised and received at least one dose of treatment (1 patient was not randomised or dosed and a further 1 patient was randomised but not dosed due to Incorrect enrolmentCediranib)
Arm/Group | Cediranib 45 mg/Day GIST | Cediranib 45 mg/Day STS
Serious Adverse Events (participants affected / at risk) | 10/24 | 3/10
Other Adverse Events (participants affected / at risk) | 24/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg/Day GIST (N=24) | Cediranib 45 mg/Day STS (N=10)
Anaemia (Vascular disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg/Day GIST (N=24) | Cediranib 45 mg/Day STS (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 2
Splinter Haemorrhages (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 20 | 8
Constipation (Gastrointestinal disorders) | 9 | 2
Nausea (Gastrointestinal disorders) | 7 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 4
Abdominal Pain (Gastrointestinal disorders) | 5 | 3
Oral Pain (Gastrointestinal disorders) | 5 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 1
Abdominal Distension (Gastrointestinal disorders) | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Mouth Ulceration (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 2
Glossodynia (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 17 | 7
Oedema Peripheral (General disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 4
Mucosal Inflammation (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 0
Furuncle (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Viral Infection (Infections and infestations) | 0 | 2
Gastric Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Tooth Infection (Infections and infestations) | 1 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Weight Decreased (Investigations) | 6 | 2
Transaminases Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 13 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 8 | 3
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Ageusia (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 2 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 19 | 4
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.